CLINICAL TRIAL: NCT01192282
Title: Clinico-Pathological HPV DNA Typing Study of Women With Genital Warts Presenting to Groote Schuur Hospital Over a One Year Period, Evaluated by HIV Status, Psychological Impact and Costs to the Health Care System
Brief Title: Typing of Human Papilloma Virus (HPV) From Female Genital Warts
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Shahila Tayib, Dr, University of Cape Town
Other Study IDs: 131/2010
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Genital Warts; Human Papilloma Virus
Keywords: Female Genital Warts; HPV Typing; HIV Status; Treatment Modalities and Recurrence; Socio-economic Burdens
MeSH Terms: conditions — Condylomata Acuminata; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genital Warts: All female patients with Genital Warts presenting to Groote Schuur Hospital
  Interventions: Procedure: Medical / Surgical Treatment

INTERVENTIONS:
Procedure: Medical / Surgical Treatment — All participants received treatment based on the morphology and distributions of lesions. For the treatment with Trichloroacetic Acid (TCA), patients were advised to attend the clinic weekly until no visible lesions seen. For electrosurgery or laser, patients were given a date for admission a day prior to surgery. Post-operatively, she remained in the ward for at least five days.

SUMMARY:
This is a longitudinal observational study of women presenting to Groote Schuur Hospital with genital warts. The study will evaluate the socio-demographic characteristics of the women using a structured questionnaire. It will also document the site and extend of the genital warts and genotyping will be performed on the warts. HIV status will be determined with patient consent, treatment modalities will be documented as will the outcome of treatment over a 6 month's period. Risk factors for recurrence or failure of treatment will be analysed as will the costs of treating women with genital warts.

DETAILED DESCRIPTION:
Genital Human Papillomavirus (HPV) infection is the most common sexually transmitted viral disease in the world.1,2 HPV infection on genital epithelia is associated with a range of disease spectra, from visible lesions such as genital warts, cervical, vaginal, vulval, anal and penile intraepithelial cancers and their precursors, or they may co- exist in the latent form in apparently normal epithelium.3,4 It is established that genital warts are associated with low-risk HPV genotypes, with the causative agents being HPV-6 and HPV-11 in almost 100% of cases.5 However, recent studies have shown that 20 to 50% of lesions also contain co-infection with high-risk HPV types.6,7

Although genital warts are not life-threatening, they cause significant psychosocial morbidities resulting in low self-esteem, negative self-perception, embarrassment and anxiety.8,9 Genital warts also represent not only a health problem for the individual, but also an economic burden for society as they carry a high and immediate financial burden and health care cost due to their generally recalcitrant response to conventional therapies.9 With this in mind, immunization with HPV 6/11/16/18 recombinant vaccine holds promise for reducing overall burden on clinical HPV-related diseases.

Genital warts are a common cause for referral to the Colposcopy Clinic of Groote Schuur Hospital, Cape Town which is a tertiary hospital serving the wider Cape Town area and the Western Cape Province. With an increasing number of cases seen requiring multiple clinical visits for treatment and a high number of recurrent and persistent cases, we undertook this study to examine the nature of the disease from a clinical point of view, response to various therapies, the impact of HIV and the types of HPV causing or associated with genital warts in women referred to our clinic.

ELIGIBILITY:
Inclusion Criteria:

* All female patients with genital warts

Exclusion Criteria:

* Patients who are pregnant, too frail or ill for gynaeoclogical examination and refusal to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All female patients with Genital Warts presenting to Groote Schuur Hospital, Cape Town
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahila Tayib, MBChB, Principal Investigator — University of Cape Town; Lynette Denny, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All female patients with genital warts referred to the Colposcopy Clinic of Groote Schuur Hospital, Cape Town, South Africa between 1st April 2010 and 30 September 2010. Those who were pregnant or too frail or ill for a gynaecological examination were excluded.
Pre-assignment Details: No Applicable.
Groups:
- Number of Participants: Participants with Genital Warts
Period: Overall Study
Arm/Group | Number of Participants
Started | 156
Completed | 156
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- New Cases: Newly diagnosed cases of genital warts
- Recurrent Cases: Reappearance of genital warts at 3 or 6 months post-treatment in participants free of warts at completion of treatment
- Persistent Cases: The warts presence after completion of treatment
- Total: Total of all reporting groups
Arm/Group | New Cases | Recurrent Cases | Persistent Cases | Total
Number analyzed (Participants) | 94 | 40 | 22 | 156
Age, Customized [Mean (Full Range); unit: Years] | 28.64 [15 to 53] | 30.18 [18 to 49] | 29.91 [17 to 50] | 29.21 [15 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 40 | 22 | 156
  Male | 0 | 0 | 0 | 0
Marital Status [Number; unit: Participants]
  Single, Not Sexually Active | 19 | 6 | 5 | 30
  Single, Sexually Active | 56 | 27 | 9 | 92
  Married | 13 | 4 | 4 | 21
  Separated / Divorced / Widow | 6 | 3 | 4 | 13
Age at First Sexual Intercourse [Number; unit: Participants]
  14 or Less (Years) | 9 | 2 | 1 | 12
  15 - 19 (Years) | 69 | 33 | 14 | 116
  20 and Above (Years) | 16 | 5 | 6 | 27
  Virgo Intacta (Years) | 0 | 0 | 1 | 1
Education Level [Number; unit: Participants]
  Primary | 13 | 0 | 3 | 16
  Secondary | 67 | 36 | 13 | 116
  Tertiary | 14 | 4 | 6 | 24
Smoking [Number; unit: Participants]
  Yes | 9 | 3 | 4 | 16
  No | 77 | 34 | 15 | 126
  Previously | 8 | 3 | 3 | 14
HIV Status [Number; unit: Participants]
  Positive | 71 | 36 | 16 | 123
  Negative | 21 | 3 | 5 | 29
  Unknown | 2 | 1 | 1 | 4
Treatment Modalities [Number; unit: Participants]
  Local Ablation with Tricholoroacetic Acid (TCA) | 7 | 2 | 2 | 11
  Electrocautery under LA | 68 | 28 | 13 | 109
  Electrocautery / Laser Ablation under GA | 17 | 9 | 7 | 33
  TCA + Electrocautery | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: HPV DNA and HIV Status
Description: HPV DNA Positivity and HIV Status
Time Frame: 18 Months
Population: Only 126 out of 156 samples collected from each patients were analysed as 30 of the samples were contaminated, of which 22 were from HIV Positive patients and 8 were from HIV Negative patients.
Measure: Number; unit: participants
Groups:
- HIV Positive: Number of participants with HIV Positive
- HIV Negative: Number of participants with HIV Negative
- HIV Unknown: Number of participants who refused HIV Testing
Arm/Group | HIV Positive | HIV Negative | HIV Unknown
Number analyzed (Participants) | 101 | 21 | 4
participants
  HPV Positive | 96 | 19 | 4
  HPV Negative | 5 | 2 | 0

2. Primary Outcome: HPV DNA and Pap Smear Results
Description: Relationship between HPV DNA Positivity and Pap Smear Results
Time Frame: 18 Months
Population: Only 118 out of 119 patients with HPV DNA Positive had a Pap Smear done. One patient was a Virgin and hence no Pap Smear was done.
Measure: Number; unit: Participants
Groups:
- HPV DNA Positive: Participants with HPV DNA Positive
- HPV DNA Negative: Participants with HPV DNA Negative
Arm/Group | HPV DNA Positive | HPV DNA Negative
Number analyzed (Participants) | 118 | 7
Participants
  Normal | 42 | 5
  Low Grade Squamous Intraepithelial Lesion | 59 | 2
  High Grade Squamous Intraepithelial Lesion | 10 | 0
  Atypical Squamous Cell of Undetermined Significanc | 6 | 0

3. Primary Outcome: Number of HPV Genotypes Isolated by HIV Status
Description: Number of HPV Genotypes isolated according to HIV Status
Time Frame: Up to 18 months
Population: 119 out of 126 uncontaminated samples were HPV DNA Positive. Out of these 119 HPV DNA Positive Samples, 12 were B-Globin Positive but no specific HPV Genotype could be identifiable.
Measure: Number; unit: participants
Groups:
- HIV Positive: Participants with HIV Positive
- HIV Negative: Participants with HIV Negative
- HIV Unknown: Participants who Refused HIV Testing
Arm/Group | HIV Positive | HIV Negative | HIV Unknown
Number analyzed (Participants) | 96 | 19 | 4
participants
  1 HPV Genotype | 44 | 14 | 1
  2 HPV Genotype | 12 | 1 | 2
  3 HPV Genotype | 9 | 2 | 0
  4 HPV Genotype | 4 | 0 | 0
  5 HPV Genotype | 5 | 0 | 0
  6 HPV Genotype | 3 | 0 | 0
  7 HPV Genotype | 5 | 0 | 0
  8 HPV Genotype | 1 | 0 | 0
  9 HPV Genotype | 1 | 0 | 0
  11 HPV Genotype | 2 | 0 | 0
  15 HPV Genotype | 1 | 0 | 0
  No Genotype Isolated but B-Globin Positive | 9 | 2 | 1

4. Primary Outcome: Commonest HPV Genotypes Isolated by HIV Status
Description: 10 commonest types of HPV isolated according to HIV status
Time Frame: 18 months
Measure: Number; unit: Participants
Arm/Group | HIV Positive | HIV Negative
Number analyzed (Participants) | 101 | 21
Participants
  HPV 11 | 46 | 10
  HPV 6 | 33 | 9
  HPV 89 | 19 | 0
  HPV 61 | 16 | 0
  HPV 55 | 12 | 0
  HPV 62 | 12 | 0
  HPV 81 | 9 | 0
  HPV 16 | 8 | 0
  HPV 18 | 8 | 0
  HPV 45 | 8 | 0

ADVERSE EVENTS:
Time Frame: 1 year and 10 months
Description: Adverse event here referred to developement of warts recurrent after treatment.
Groups:
- HIV Positive: Participants with Genital Warts who were HIV Positive
- HIV Negative: Participants with Genital Warts who were HIV Negative
- HIV Unknown: Participants with Genital Warts whom HIV Status was Unknown
Arm/Group | HIV Positive | HIV Negative | HIV Unknown
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/29 | 0/4
Other Adverse Events (participants affected / at risk) | 28/123 | 5/29 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Positive (N=123) | HIV Negative (N=29) | HIV Unknown (N=4)
Warts Recurrence (Skin and subcutaneous tissue disorders) | 28 (28) | 5 (5) | 0 (0) — Patients recruited were seen at 3 and 6 months post-treatmeant to assess warts recurrence.

LIMITATIONS AND CAVEATS:
Thirty (19.2%) specimens had to be rejected due to contamination that occurred during the analysis process. During the HPV DNA analysis, there were protocols for different aspect of controls during the analysis which needed to be negative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No